CLINICAL TRIAL: NCT01105312
Title: Phase I/II Study of Panobinostat (LBH589) and Letrozole in Patients With Triple Negative Metastatic Breast Cancer
Brief Title: Panobinostat and Letrozole in Treating Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N093B; NCCTG-N093B; CDR0000669300 (Registry Identifier: PDQ (Physician Data Query)); NCI-2011-02035 (Registry Identifier: CTRP (Clinical Trials Reporting System))
Record Dates: First submitted 2010-04-15; First posted 2010-04-16 (Estimated); Results first posted 2017-06-27 (Actual); Last update posted 2017-06-27 (Actual); Status verified 2017-05

CONDITIONS: Breast Cancer
Keywords: male breast cancer; estrogen receptor-negative breast cancer; estrogen receptor-positive breast cancer; HER2-negative breast cancer; HER2-positive breast cancer; progesterone receptor-negative breast cancer; progesterone receptor-positive breast cancer; triple-negative breast cancer; recurrent breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male; Triple Negative Breast Neoplasms | interventions — Letrozole; Panobinostat; Microarray Analysis; Reverse Transcriptase Polymerase Chain Reaction; Enzyme-Linked Immunosorbent Assay; Immunohistochemistry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- panobinostat (LBH589) and letrozole (Experimental): Each patient will receive panobinostat (LBH589) and letrozole. Patients will be administered LBH589 PO, 3 days per week for a total of 4 weeks. Patients will also be administered letrozole 2.5 mg PO Days 1-28 every 4 weeks. There are two phases of the study. The first phase determines the maximum tolerated dose for LBH589 in combination with letrozole. The second phase is to assess and confirm the response rate and safety profile of LBH589 in combination with letrozole.
  Interventions: Drug: letrozole; Drug: panobinostat; Genetic: RNA analysis; Genetic: microarray analysis; Genetic: reverse transcriptase-polymerase chain reaction; Other: enzyme-linked immunosorbent assay; Other: immunohistochemistry staining method; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: letrozole
Drug: panobinostat
Genetic: RNA analysis
Genetic: microarray analysis
Genetic: reverse transcriptase-polymerase chain reaction
Other: enzyme-linked immunosorbent assay
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Panobinostat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Estrogen can cause the growth of breast cancer cells. Hormone therapy using letrozole may fight breast cancer by lowering the amount of estrogen the body makes. Giving panobinostat together with letrozole may be an effective treatment for breast cancer.

PURPOSE: This phase I/II trial is studying the side effects and best dose of panobinostat when given together with letrozole and to see how well it works in treating patients with metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary Objectives

* To determine the maximum-tolerated dose of panobinostat in combination with letrozole in patients with metastatic breast cancer. (Phase I)
* To determine the safety of this regimen in these patients. (Phase I)
* To assess the confirmed response rate and safety profile of this regimen in patients with triple-negative disease. (Phase II)

Secondary Objectives

* To assess the therapeutic effects of this regimen in these patients. (Phase I)
* To examine the duration of response, clinical benefit rate, and time to treatment failure in patients treated with this regimen. (Phase II)
* To examine the time to progression, progression-free survival, and overall survival of patients treated with this regimen. (Phase II)
* To examine the estrogen, progesterone, and HER2 status of tumor at primary compared to metastatic tissue, and possibly after treatment. (exploratory)
* To bank paraffin-embedded tissue blocks/slides and blood products for future studies. (exploratory)
* To determine expression levels of biomarkers of treatment response (i.e., ER, PR, aromatase, NFkappaB, Ki67, and Caspase 3) in accessible tumors pre- and post-therapy via immunohistochemistry. (exploratory)
* To determine whether ELISA for KLK11 in serum can be used as marker of activity of letrozole and LBH589. (exploratory) The Phase I portion of this study closed and the Phase II portion of the study opened as per NCCTG Addendum 6, effective January 23, 2012.

OUTLINE: This is a multicenter, phase I dose-escalation study of panobinostat followed by a phase II study. (The Phase I portion of this study closed and the Phase II portion of the study opened as per NCCTG Addendum 6, effective January 23, 2012.)

Patients receive oral panobinostat once daily on days 1, 3, and 5 in weeks 1-4 and oral letrozole once daily on days 1-28. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

Tumor tissue and blood samples are collected and banked for future biomarker and other analysis. Samples are also analyzed for biomarkers utilizing immunohistochemistry, microarray, reverse transcription-polymerase chain reaction (RT-PCR), and enzyme-linked immunosorbent assay (ELISA).

After completion of study therapy, patients are followed up every 3-6 months for up to 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed breast cancer

  * Metastatic disease amenable to biopsy
  * Unresected tumor with no intention to undergo resection during study
* Archival tissue from the primary diagnosis or fresh biopsy from metastatic cancer site required
* Measurable or non-measurable disease for phase I study (The Phase I portion of this study closed and the Phase II portion of the study opened as per NCCTG Addendum 6, effective January 23, 2012.)

  * Measurable disease only for phase II study
* Available tumor estrogen (ER), progesterone (PR), and HER2 status from metastatic site tested by IHC or FISH OR results from the original tumor diagnosis

  * Any ER, PR, or HER2 level (positive or negative) acceptable (phase I)
  * Triple-negative disease only (phase II)

    * ER and PR negative defined as ≤ 1% by IHC
    * HER2 negative

      * Patients with triple-negative breast cancer allowed provided there is clinical or radiographic evidence of tumor progression in the adjuvant or metastatic setting
* No patients whose disease can be treated with known standard therapy that is potentially curative or definitely capable of extending life expectancy
* No known CNS metastasis
* Hormone-receptor status:

  * ER and PR positive or negative (phase I)
  * ER and PR negative (phase II)

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1 (phase I) or 0-2 (phase II)
* Postmenopausal defined by 1 of the following:

  * ≥ 60 years of age
  * ≥ 45 years of age with last menstrual period ≥ 12 months prior and estradiol and follicle-stimulating hormone levels in postmenopausal range
  * Bilateral oophorectomy
* Life expectancy ≥ 12 weeks
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Total bilirubin normal
* ALT and AST ≤ 3 times upper limit of normal (ULN) (≤ 5 times ULN if due to liver metastasis)
* Serum creatinine ≤ 1.5 times ULN
* TSH normal (thyroid hormone supplements allowed for patients with hypothyroidism)
* Not pregnant or nursing
* Fertile patients must use effective contraception
* Willing to return to Mayo Clinic or NCCTG institution (phase II) for follow-up
* Willing to provide blood samples for correlative research purposes
* No uncontrolled or intercurrent illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness and/or social situations that would limit compliance with study requirements
* No NYHA class III or IV cardiovascular disease
* No known seizure disorder
* No co-morbid systemic illnesses or other severe concurrent disease that, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* No immunocompromised patients, including patients known to be HIV positive

  * Immunocompromised patients due to the use of corticosteroids allowed
* No malignancy within the past 5 years except for nonmelanoma skin cancer or carcinoma in situ of the cervix
* No history of myocardial infarction ≤ 6 months
* No congenital long QT syndrome or QTcF>450 msec, including:

  * Complete left bundle block or use of a permanent cardiac pacemaker, history or presence of ventricular tachyarrhythmias, clinically significant resting bradycardia (<50 beats per minute)
  * Right bundle branch block + left anterior hemiblock (bifascicular block)
* No congestive heart failure requiring use of maintenance therapy for life-threatening ventricular arrhythmias

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 4 weeks since prior chemotherapy or radiotherapy and fully recovered

  * No radiotherapy to > 25 % of bone marrow
* Prior treatments allowed (phase II):

  * 0 or 1 prior chemotherapy regimens for breast cancer
  * ≤ 2 prior aromatase-inhibitor regimens (including letrozole)
* Not currently receiving treatment in a different clinical study in which investigational procedures are performed or investigational therapies are administered
* No other concurrent investigational agent for the primary neoplasm
* No concurrent CYP3A4 inhibitors or inducers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-09 (Actual); Primary Completion 2013-08 (Actual); Study Completion 2013-09-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Winston Tan, MD, FACP, Study Chair — Mayo Clinic
Locations (172):
- United States (172):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Contra Costa Regional Medical Center, Martinez, California
  - El Camino Hospital Cancer Center, Mountain View, California
  - Bay Area Breast Surgeons, Incorporated, Oakland, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Larry G Strieff MD Medical Corporation, Oakland, California
  - Tom K Lee, Incorporated, Oakland, California
  - Pismo Beach, California
  - Doctors Medical Center - San Pablo Campus, San Pablo, California
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - St. Anthony Central Hospital, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - St. Mary - Corwin Regional Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Florida Hospital Memorial Medical Center, Daytona Beach, Florida
  - Michael and Dianne Bienes Comprehensive Cancer Center at Holy Cross Hospital, Fort Lauderdale, Florida
  - Memorial Cancer Institute at Memorial Regional Hospital, Hollywood, Florida
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Ella Milbank Foshay Cancer Center at Jupiter Medical Center, Jupiter, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - John B. Amos Cancer Center, Columbus, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Lusitana, Honolulu, Hawaii
  - Queen's Cancer Institute at Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Incorporated, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Kuakini, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Kauai Medical Clinic, Lihue, Hawaii
  - Kapiolani Medical Center at Pali Momi, ‘Aiea, Hawaii
  - Oncare Hawaii, Incorporated - Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center at Saint Alphonsus Regional Medical Center, Boise, Idaho
  - Illinois CancerCare - Bloomington, Bloomington, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare - Canton, Canton, Illinois
  - Illinois CancerCare - Carthage, Carthage, Illinois
  - Resurrection Medical Center, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Illinois CancerCare - Eureka, Eureka, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Illinois CancerCare - Havana, Havana, Illinois
  - Illinois CancerCare - Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare - Macomb, Macomb, Illinois
  - Illinois CancerCare - Monmouth, Monmouth, Illinois
  - OSF Holy Family Medical Center, Monmouth, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Illinois CancerCare - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Illinois CancerCare - Pekin, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare - Peru, Peru, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Illinois CancerCare - Princeton, Princeton, Illinois
  - Illinois CancerCare - Spring Valley, Spring Valley, Illinois
  - McFarland Clinic, PC, Ames, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas, PA - Liberal, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Alvin and Lois Lapidus Cancer Institute at Sinai Hospital, Baltimore, Maryland
  - Peninsula Regional Medical Center, Salisbury, Maryland
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - CCOP - Hematology-Oncology Associates of Central New York, East Syracuse, New York
  - Monter Cancer Center of the North Shore-LIJ Health System, Lake Success, New York
  - Don Monti Comprehensive Cancer Center at North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Moses Cone Regional Cancer Center at Wesley Long Community Hospital, Greensboro, North Carolina
  - Pardee Memorial Hospital, Hendersonville, North Carolina
  - Kinston Medical Specialists, Kinston, North Carolina
  - Annie Penn Cancer Center, Reidsville, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - Altru Cancer Center at Altru Hospital, Grand Forks, North Dakota
  - Wood County Oncology Center, Bowling Green, Ohio
  - Community Cancer Center, Elyria, Ohio
  - Hematology Oncology Center, Elyria, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - St. Anne Mercy Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Geisinger Hazleton Cancer Center, Hazleton, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - Oncology Services of Aberdeen, Aberdeen, South Dakota
  - Danville Regional Medical Center, Danville, Virginia
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Gundersen Lutheran Center for Cancer and Blood, La Crosse, Wisconsin
  - Holy Family Memorial Medical Center Cancer Care Center, Manitowoc, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - St. Nicholas Hospital, Sheboygan, Wisconsin

REFERENCES:
- [Derived] Tan WW, Allred JB, Moreno-Aspitia A, Northfelt DW, Ingle JN, Goetz MP, Perez EA. Phase I Study of Panobinostat (LBH589) and Letrozole in Postmenopausal Metastatic Breast Cancer Patients. Clin Breast Cancer. 2016 Apr;16(2):82-6. doi: 10.1016/j.clbc.2015.11.003. Epub 2015 Nov 17. PMID 26774555

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase II; Phase I: Dose Level One: Each patient will receive panobinostat (LBH589) and letrozole. Patients will be administered 20 mg LBH589 PO, 3 days per week for a total of 4 weeks. Patients will also be administered letrozole 2.5 mg PO Days 1-28 every 4 weeks.
- Phase I: Dose Level Two: Each patient will receive panobinostat (LBH589) and letrozole. Patients will be administered 30 mg LBH589 PO, 3 days per week for a total of 4 weeks. Patients will also be administered letrozole 2.5 mg PO Days 1-28 every 4 weeks.
Period: Overall Study
Arm/Group | Phase II | Phase I: Dose Level One | Phase I: Dose Level Two
Started | 16 | 6 | 6
Completed | 13 | 6 | 6
Not Completed | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All phase I and phase II patients were used for baseline analysis
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase II | Phase I: Dose Level One | Phase I: Dose Level Two | Total
Number analyzed (Participants) | 16 | 6 | 6 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 3 | 4 | 18
  >=65 years | 5 | 3 | 2 | 10
Age, Continuous [Median (Full Range); unit: years] | 60.5 [43 to 75] | 66 [56 to 75] | 63 [43 to 68] | 62.5 [43 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 6 | 6 | 28
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 6 | 6 | 28

OUTCOME MEASURES:

1. Primary Outcome: Maximum-tolerated Dose (Phase I)
Description: MTD is defined as the dose level below the lowest dose that induces dose limiting toxicity in at least one-third of patients (at least 2 of a maximum of 6> new patients). If dose-limiting toxicity (DLT) is not seen in any of the 3 patients, 3 new patients will be accrued and treated at the next higher dose level. If DLT are seen in 2 or 3 of 3 patients treated at a given dose level, then the next 3 patients will be treated at the next lower dose level, if only 3 patients were enrolled and treated at this lower dose level. The number of DLT's will be reported here.
Time Frame: Up to 2.5 months
Population: All 12 phase I patients were eligible and analyzed for MTD.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: Dose Level One | Phase I: Dose Level Two
Number analyzed (Participants) | 6 | 6
Participants | 1 | 3

2. Primary Outcome: Response Rate (Phase II)
Description: A confirmed response is defined to be a CR or PR (as determined by RECIST (version 1.1 criteria) noted as the objective status on 2 consecutive evaluations at least 4 weeks apart. Response will be evaluated using all cycles of treatment. All patients meeting the eligibility criteria who have signed a consent form and have begun treatment will be evaluable for response.
  A CR is defined as:
  All of the following must be true:
  1. Disappearance of all non-nodal target lesions
  2. Each target lymph node must have reduction in short axis to <1.0 cm
  A PR is defined as:
  At least a 30% decrease in the sum of the longest diameters of the non-nodal target lesions and the short axes of the target lymph nodes taking as reference the BSD (Section 11.41)
Time Frame: from baseline up to 5 years post-registration
Population: 13 of the 16 patients enrolled were eligible, treated, and analyzed for this endpoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase II
Number analyzed (Participants) | 13
percentage of participants | 0 [0 to 24.7]

3. Secondary Outcome: Survival Time (Phase II)
Description: Survival time is defined as the time from registration to death due to any cause. The distribution of survival time will be estimated using the method of Kaplan-Meier
Time Frame: from baseline up to 5 years post-registration
Population: 13 of the 16 phase II patients were eligible, treated, and analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II
Number analyzed (Participants) | 13
months | 16.1 [13.4 to NA] — The data is skewed due to small sample size (insufficient number of participants with events)

4. Secondary Outcome: Time-to-disease Progression (Phase II)
Description: Time-to-disease progression (TTP) is defined as the time from registration to documentation of disease progression. If a patient dies without a documentation of disease progression, the patient will be considered to have had tumor progression at the time of their death unless there is sufficient documented evidence to conclude no progression occurred prior to death. The distribution of TTP will be estimated using the method of Kaplan-Meier. Progression is defined as at least one of the following:
  1. At least one new malignant lesion or a lymph node whose short axis has increased to >1.5 cm
  2. At least a 20% increase in the sum of diameters of target lesions taking as reference the MSD. In addition, the sum must also demonstrate an absolute increase of at least 0.5 cm
Time Frame: from baseline up to 6 months
Population: 13 of the 16 phase II patients were eligible, treated, and analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II
Number analyzed (Participants) | 13
months | 2.1 [1.5 to NA] — The data is skewed due to small sample size (insufficient number of participants with events)

5. Secondary Outcome: Progression-free Survival (Phase II)
Description: Progression-free survival (PFS) is defined as the time from registration to progression or death due to any cause. PFS at 6 months will be estimated. The distribution of PFS will be estimated using the method of Kaplan-Meier.
Time Frame: from baseline up to 6 months
Population: 13 of the 16 phase II patients were eligible, treated, and analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II
Number analyzed (Participants) | 13
months | 2.1 [1.5 to NA] — The data is skewed due to small sample size (insufficient number of participants with events)

6. Secondary Outcome: Duration of Response (Phase II)
Description: Duration of response is defined for all evaluable patients who have achieved a confirmed response as the date at which the patient's objective status is first noted to be a CR or PR to the earliest date progression is documented. The distribution of duration of response will be estimated using the method of Kaplan-Meier.
Time Frame: from baseline up to 5 years post-registration
Population: 13 of the 16 phase II patients were treated and analyzed
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II
Number analyzed (Participants) | 13
months | NA [NA to NA] — There were no responders and thus no data to assess this endpoint.

7. Secondary Outcome: Clinical Benefit Rate
Description: Clinical benefit rate will be estimated by the total number of patients with an objective status of CR, PR, or SD for duration of at least 6 months divided by the total number of evaluable patients. All evaluable patients will be used for this analysis. Exact binomial 95% confidence intervals for the true clinical benefit rate will be calculated.
Time Frame: from baseline up to 6 months
Population: 13 of the 16 phase II patients were eligible, treated, and analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase II
Number analyzed (Participants) | 13
percentage of participants | 0 [0 to 24.7]

8. Secondary Outcome: Time to Treatment Failure
Description: Time to treatment failure (TTF) is defined as the time from the date of registration to the date at which the patient is removed from treatment due to progression, unacceptable adverse events, or refusal. The distribution of TTF will be estimated using the method of Kaplan-Meier
Time Frame: from baseline up to 5 years post-registration
Population: 13 of the 16 phase II patients were eligible, treated, and analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II
Number analyzed (Participants) | 13
months | 2 [1.1 to NA] — The data is skewed due to small sample size (insufficient number of participants with events)

9. Secondary Outcome: Confirmed Response Rate (Phase I)
Description: A confirmed response is defined to be a CR or PR (as determined by RECIST criteria) noted as the objective status on 2 consecutive evaluations at least 4 weeks apart. Response will be evaluated using all cycles of treatment. All patients meeting the eligibility criteria who have signed a consent form and have begun treatment will be evaluable for response. The number of confirmed responses will be reported here.
Time Frame: from baseline up to 5 years
Population: All 12 eligible phase I patients were treated and analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: Dose Level One | Phase I: Dose Level Two
Number analyzed (Participants) | 6 | 6
Participants | 0 | 2

ADVERSE EVENTS:
Arm/Group | Phase II | Phase I: Dose Level One | Phase I: Dose Level Two
Serious Adverse Events (participants affected / at risk) | 4/16 | 1/6 | 2/6
Other Adverse Events (participants affected / at risk) | 13/16 | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase II (N=16) | Phase I: Dose Level One (N=6) | Phase I: Dose Level Two (N=6)
Bladder infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 3 (3) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase II (N=16) | Phase I: Dose Level One (N=6) | Phase I: Dose Level Two (N=6)
Anemia (Blood and lymphatic system disorders) | 9 (15) | 4 (12) | 2 (2)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2)
Nausea (Gastrointestinal disorders) | 2 (3) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (5) | 1 (1) | 2 (6)
Bladder infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 2 (2)
Creatinine increased (Investigations) | 5 (12) | 3 (5) | 4 (9)
Electrocardiogram QT corrected interval prolonged (Investigations) | 5 (6) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 4 (8) | 3 (7) | 6 (9)
Platelet count decreased (Investigations) | 9 (15) | 5 (18) | 6 (20)
Weight loss (Investigations) | 1 (3) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 5 (9) | 5 (15) | 4 (5)
Anorexia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 1 (1)
Glucose intolerance (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2)
Hypermagnesemia (Metabolism and nutrition disorders) | 2 (2) | 3 (5) | 2 (5)
Hypocalcemia (Metabolism and nutrition disorders) | 6 (8) | 2 (7) | 4 (9)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less